CLINICAL TRIAL: NCT04524416
Title: A Prospective, Open, Multicentre Study Analysing the Long-term Safety of MINIject Glaucoma Implants in Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications
Brief Title: MINIject Global Long-Term Follow-up Study
Acronym: STAR-GLOBAL
Status: Recruiting | Type: Observational
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: STAR-GLOBAL (ISM09)
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Intra Ocular Pressure (IOP) reduction; Glaucoma Drainage Device; Minimally Invasive Glaucoma Surgery (MIGS); Supraciliary space; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Minimally invasive glaucoma surgery (MIGS) — MINIject implant placed into supraciliary space. The implantation was done in a previous study in which patient participated and is not part of this study.

SUMMARY:
The study will assess the long-term (up to 5 years) safety and performance in patients with open-angle glaucoma uncontrolled by topical hypotensive medications who had previously been implanted with a MINIject glaucoma implant.

DETAILED DESCRIPTION:
The study aims to assess long-term safety and performance of MINIject glaucoma implant up to 5 years post-implantation. Patients who received implant and were followed for 2 years in a previous study, will be invited to continue long-term follow-up from 2 to 5 years post-implantation at annual intervals. Standard ophthalmologic assessments including measurement of intraocular pressure, fundus examination, ocular imaging, assessment of any untoward ocular events etc. will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received a MINIject glaucoma implant within a prior clinical study
* Patient continues to have MINIject implanted at the point of enrolment
* Patient must provide written informed consent to participate

Exclusion Criteria:

* Individuals under tutorship or trusteeship
* Patient who is unwilling to return to the study visits and undergo study assessments, as required by clinical study protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with open-angle glaucoma not-controlled with hypotensive medications and who, to treat this condition, already received MINIject in a previous study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with serious device-related adverse event in study eye | 5 years post-implantation
  The proportion of patients with at least one serious ocular adverse event in the study eye, related to the device, occurring between 2 and 5 years after the MINIject implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — iSTAR Medical
Locations (9):
- Clinica Oftalmologica del Caribe, Barranquilla, Colombia
- France (2):
  - Center Hospotalier Universitaire Genoble Alpes, Grenoble
  - Hopital de la Croix-Rousse, Lyon
- Germany (3):
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Mainz, Mainz, Rhineland-Palatinate
  - Klinikum der Universität München, München
- Maxivision Eye Hospital, Hyderabad, Telangana, India
- Panama Eye Center, Panama City, Panama
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No